CLINICAL TRIAL: NCT05310266
Title: Ultrasound-guided Transversus Abdominis Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Laparoscopic Appendectomy: A Prospective, Randomized, Controlled Clinical Study
Brief Title: Transversus Abdominis Plane Block Versus Quadratus Lumborum Block for Pain Management in Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Gokhan Sertcakacilar, MD, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2020-35
Record Dates: First submitted 2022-03-26; First posted 2022-04-04 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain; Appendicitis Acute; Surgery
Keywords: Postoperative pain; Laparoscopic appendectomy; Transversus abdominis plane block; Quadratus Lumborum Block; Local anesthetic
MeSH Terms: conditions — Pain, Postoperative; Appendicitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TAP (Active Comparator): The investigators performed transversus abdominis plane block to that patient group for postoperative analgesia
  Interventions: Procedure: Transversus abdominis plane block
- Group QLB (Active Comparator): The investigators performed quadratus lumborum block to that patient group for postoperative analgesia
  Interventions: Procedure: Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Transversus abdominis plane block — The investigators performed transversus abdominis plane block to that patient group for postoperative analgesia
  Arms: Group TAP
Procedure: Quadratus Lumborum Block — The investigators performed quadratus lumborum block to that patient group for postoperative analgesia
  Arms: Group QLB

SUMMARY:
Laparoscopic appendectomy causes postoperative pain. The primary objective of this prospective randomized controlled study is to compare the effect of ultrasound (US)-guided quadratus lumborum block (QLB) on 24-hour cumulative opioid requirements with transversus abdominis plane (TAP) block.

DETAILED DESCRIPTION:
168 patients (ASA I-II-III) between 18 and 65 years of age, who were to undergo laparoscopic appendectomy, were randomized and divided into two groups. 32 patients were dropout for different reasons.(68 patients in each of the TAP block and QLB block groups). TAP block was performed for TAP group and QLB block was performed for QLB group. Postoperative analgesia was provided by intravenous tramadol hydrochloride using a patient-controlled analgesia device. 24-hour total tramadol hydrochloride consumption was primary outcome measure.Postoperative numeric rating scale values were the secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-65
* Patients who will undergo laparoscopic appendectomy
* ASA I-II-III patients

Exclusion Criteria:

* Clinically known local anesthetic allergy
* Morbid obesity (body mass index>40 kg m2)
* Clinically diagnosis of opioid, alcohol and substance dependence
* Clinically diagnosis of psychiatric disease
* Coagulopathy
* Patients with ASA IV-V

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Postoperative 24-hours total tramadol hydrochloride consumption | 24 hours postoperatively
  This will be measured by pca device in the 24 hour after

SECONDARY OUTCOMES:
Numerical rating scale (NRS) scores of patients | 24 hours postoperatively
  Numerical rating scale (NRS) at 1, 6, 12, 18, 24th hours. A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr. Sadi Konuk Research and Training Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data available from the publication date can start. NRS scores will be shared. If requested, data will be shared with anesthesiologists dealing with postoperative pain management.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year within the publication date.

REFERENCES:
- [Result] Tupper-Carey DA, Fathil SM, Tan YK, Kan YM, Cheong CY, Siddiqui FJ, Assam PN. A randomised controlled trial investigating the analgesic efficacy of transversus abdominis plane block for adult laparoscopic appendicectomy. Singapore Med J. 2017 Aug;58(8):481-487. doi: 10.11622/smedj.2016068. Epub 2016 Apr 8. PMID 27056207
- [Result] Baytar C, Yilmaz C, Karasu D, Topal S. Comparison of Ultrasound-Guided Subcostal Transversus Abdominis Plane Block and Quadratus Lumborum Block in Laparoscopic Cholecystectomy: A Prospective, Randomized, Controlled Clinical Study. Pain Res Manag. 2019 Feb 3;2019:2815301. doi: 10.1155/2019/2815301. eCollection 2019. PMID 30863471
- [Result] Saleh AH, Abdallah MW, Mahrous AM, Ali NA. Quadratus lumborum block (transmuscular approach) versus transversus abdominis plane block (unilateral subcostal approach) for perioperative analgesia in patients undergoing open nephrectomy: a randomized, double-blinded, controlled trial. Braz J Anesthesiol. 2021 Jul-Aug;71(4):367-375. doi: 10.1016/j.bjane.2021.01.009. Epub 2021 Mar 21. PMID 33762197